CLINICAL TRIAL: NCT01465113
Title: Effect of Vitamin D Supplementation on 15-Prostaglandin Dehydrogenase Expression in Barrett's Esophagus
Brief Title: Vitamin D Supplementation on 15-Prostaglandin Dehydrogenase Expression in Barrett's Esophagus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASE12209
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Short Segment Barrett's Esophagus; Long Segment Barrett's Esophagus
Keywords: Barrett's Esophagus; Vitamin D3; cholecalciferol; 15-Prostaglandin Dehydrogenase Expression; metformin
MeSH Terms: conditions — Barrett Esophagus | interventions — Omeprazole; Cholecalciferol; Gastroscopy; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Indefinite, LGD or no dysplasia arm (Experimental): Barrett's esophagus patients who have no dysplasia or low grade dysplasia
  Interventions: Drug: Omeprazole; Drug: Vitamin D3; Procedure: upper endoscopy
- high grade dysplasia (Experimental): Barrett's esophagus with high grade dysplasia
  Interventions: Drug: Omeprazole; Drug: Vitamin D3; Procedure: upper endoscopy
- Indefinite, LGD or no dysplasia arm:Vitamin D/Metformin Subarm (Experimental): Barrett's esophagus patients who have no dysplasia or low grade dysplasia
  Interventions: Drug: Omeprazole; Drug: Vitamin D3; Procedure: upper endoscopy; Drug: Metformin

INTERVENTIONS:
Drug: Omeprazole — 28-day run-in phase during which subjects are treated with a proton pump inhibitor (omeprazole 20 mg po q day or an equivalent dose of another proton pump inhibitor).
Drug: Vitamin D3 — These patients (indefinite for dysplasia, LGD, or no dysplasia) will take vitamin D3 50,000 IU once a week for 12 weeks following the upper endoscopy.
  Other Names: Cholecalciferol
  Arms: Indefinite, LGD or no dysplasia arm; Indefinite, LGD or no dysplasia arm:Vitamin D/Metformin Subarm
Drug: Vitamin D3 — Due to the risk of progression, subjects with Barrett's esophagus with high grade dysplasia will take vitamin D3 50,000 IU once a week for 2 weeks.
  Other Names: Cholecalciferol
  Arms: high grade dysplasia
Procedure: upper endoscopy — After the run-in phase subjects will undergo an upper endoscopy for Barrett's surveillance or Barrett's mapping as part of routine clinical care. At the time of endoscopy, in addition to large cup forceps biopsies obtained for surveillance or mapping as part of standard care, research biopsies will be obtained for the study. Following vitamin D3 supplementation, all subjects will undergo a repeat upper endoscopy for additional large cup forceps biopsies for measurement of post-treatment mucosal levels.
Drug: Metformin — 500mg for the first week, 1000mg during the second week, 1500mg during the third week, maximum dose of 2000mg in the fourth week
  Arms: Indefinite, LGD or no dysplasia arm:Vitamin D/Metformin Subarm

SUMMARY:
This study is being conducted to determine if vitamin D supplementation increases the level of a protein that may be involved in decreasing the risk of esophageal cancer in patients with Barrett's esophagus. Subjects with Barrett's esophagus will take vitamin D supplementation for 2-12 weeks depending on the severity of their condition, and receive an upper endoscopy procedure before and after vitamin D supplementation trial.

DETAILED DESCRIPTION:
28-day run-in phase during which subjects are treated with a proton pump inhibitor (omeprazole 20 mg po q day or an equivalent dose of another proton pump inhibitor). The purpose of the run-in phase is to minimize esophagitis, which can cause histologic changes that can be confused with dysplasia. After the run-in phase, subjects will undergo an upper endoscopy for Barrett's surveillance or Barrett's mapping as part of routine clinical care. At the time of endoscopy, research biopsies will be obtained for the study. Subjects eligible and continuing in the study will take vitamin D3 (Cholecalciferol) 50,000 IU capsules once weekly with or without daily metformin for a total of two or twelve weeks depending on the severity of Barrett's esophagus. After completion of vitamin D3 subjects will return for an EGD (endoscopy) and biopsies for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of short-segment or long-segment Barrett's esophagus as previously made by upper endoscopy showing salmon-colored distal esophageal mucosa and biopsies revealing intestinal metaplasia with goblet cells. Potential study subjects may be contacted by mailings or phone calls or may be approached in clinic. Additionally, potential study subjects may be approached using a web-based recruitment tool. Informed consent will be obtained by a research coordinator or study investigator.
* Subjects may be taking calcium supplements or have previous history of hypercalcemia
* Subjects may have diabetes mellitus
* Subjects may have a history of prior malignancy except for esophageal adenocarcinoma
* Willing to donate 90 mL of blood and endoscopic mucosal biopsies for research

The following additional inclusion criteria apply for patients in the Vitamin D/metformin sub-arm of the low grade dysplasia/no dysplasia arm:

* At least 2 cm circumferential Barrett's esophagus segment length (C2M2 by Prague C & M criteria)
* Normal renal function (defined as creatinine within normal institutional limits)

Exclusion Criteria:

* Pregnancy
* Known chronic liver disease (Child's B cirrhosis)
* Known chronic kidney disease (creatinine ≥ 3.0)
* Esophageal adenocarcinoma
* Allergic reaction to omeprazole
* Allergic reaction to vitamin D
* Unable or unwilling to provide informed consent
* Known hypercalcemia
* Previous ablative therapy for Barrett's esophagus
* Patients on a stable (>/=4 week duration) dose of >2000 IU/day (or equivalent) of vitamin D supplementation

The following additional exclusion criteria apply for patients in the Vitamin D/metformin sub-arm of the no dysplasia/low grade dysplasia arm:

* Allergic reaction to metformin
* History of diabetes mellitus
* History of lactic acidosis
* History of B12 deficiency
* Participants may not be using metformin, cimetidine (Tagamet) furosemide (Lasix), nifedipine (Cardizem), or any other drug contraindicated for use with metformin.
* Treatment with other oral hypoglycemic agents
* Participants planning to undergo elective radiologic studies involving intravascular administration of iodinated contrast materials.
* Known chronic kidney disease with creatinine greater than normal institutional limits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Arm 1(no or low grade dysplasia): 15-Prostaglandin dehydrogenase expression | after 12 weeks of vitamin D supplement
  To determine whether vitamin D supplementation induces 15-Prostaglandin dehydrogenase expression as measured by RT-PCR in Barrett's esophagus
Arm 2 (high grade dysplasia): 15-Prostaglandin dehydrogenase expression | after 2 weeks of vitamin D supplement
  To determine whether vitamin D supplementation induces 15-Prostaglandin dehydrogenase expression as measured by RT-PCR in Barrett's esophagus

SECONDARY OUTCOMES:
decreased prostaglandin E2 expression in Barrett's esophagus | after 2 or 12 weeks of vitamin D supplement
  To determine whether vitamin D supplementation leads to decreased prostaglandin E2 expression in Barrett's esophagus
effects on cyclooxygenase-2 expression | after 2 or 12 weeks after vitamin D supplement
  To determine whether vitamin D supplementation affects cyclooxygenase-2 expression in Barrett's esophagus
15-Prostaglandin dehydrogenase expression differences between RT-PCR and immunohistochemistry | after 2 or 12 weeks after vitamin D supplement
  To determine whether 15-Prostaglandin dehydrogenase expression in Barrett's esophagus differs between RT-PCR and immunohistochemistry
effects on levels of Ki-67 | after 2 or 12 weeks after vitamin D supplement
  To determine whether vitamin D supplementation affects levels of Ki-67, a marker for proliferation, in Barrett's esophagus
effects on levels of caspase | after 2 or 12 weeks of vitamin D supplement
  To determine whether vitamin D supplementation affects levels of caspase, a marker for apoptosis, in Barrett's esophagus
effects on insulin resistance | after 2 or 12 weeks of vitamin D supplement
  To determine whether vitamin D supplementation affects insulin resistance in Barrett's esophagus

CONTACTS AND LOCATIONS:
Overall Officials: Linda Cummings, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University Hospitals Ahuja Medical Center, Beachwood, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio